CLINICAL TRIAL: NCT01938326
Title: Postoperative Pain and Quality of Life After Single-incision Distal Gastrectomy Versus Totally Laparoscopic Distal Gastrectomy for Early Gastric Cancer - a Randomized Controlled Trial
Brief Title: Pure Single Incision Laparoscopic Distal Gastrectomy (SIDG) Versus Totally Laparoscopic Distal Gastrectomy (TLDG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Sang-Hoon Ahn, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-SIDG-GS-PII
Record Dates: First submitted 2012-07-15; First posted 2013-09-10 (Estimated); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Early Gastric Cancer
Keywords: Stomach neoplasm; TLDG; SIDG; single-port; inflammatory response
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-port laparoscopic distal gastrectomy (Active Comparator): Laparoscopic distal gastrectomy using the conventional 5-port access
  Interventions: Procedure: Approach Method
- Single incision distal gastrectomy (Active Comparator): Pure single incision distal gastrectomy using one transumbilical incision
  Interventions: Procedure: Approach Method

INTERVENTIONS:
Procedure: Approach Method — SIDG : 1 incision (umbilicus 2.5cm) TLDG : 5 incisions (12mm ports X 3, 5mm ports X 2, umbilicus extension up to 3cm for specimen delivery)

SUMMARY:
1. Compare the immune response and postoperative complications between pure SIDG (single-incision laparoscopic distal gastrectomy) and TLDG (totally laparoscopic distal gastrectomy) for early gastric cancer (EGC)
2. Validate the safety, usefulness, minimal invasiveness and feasibility of SIDG (EGC)

DETAILED DESCRIPTION:
There are some trends of reducing the numbers and lengths of wounds in the fields of laparoscopic surgery.

Recently, Beyond laparoscopy-assisted distal gastrectomy (LADG), which has the mini-laparotomy, TLDG, which has no mini-laparotomy in epigastrium but in umbilicus, has been popular procedure in the treatment of gastric cancer. Furthermore, the report on early experience of SIDG, which has no incision except umbilicus port, is going to be published.

However, there've been no objective reports and data on real minimal invasiveness and benefits between 2 procedures. In this study, I would like to find out the benefits of the reducing port and wound size by comparing the above 2 procedures' immune response and postoperative complications.

This study is planned as a phase II study.

There are no references on this subject, so the investigators set the numbers of each groups into 30, which is minimal requirement for the parametric comparisons.

ELIGIBILITY:
Inclusion Criteria:

* clinically early gastric cancer, potentially possible to perform distal gastrectomy (cancer in the distal 2/3rds)
* 20< Age < 80

Exclusion Criteria

* history of other malignancy
* received preoperative chemotherapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Maximum pain score using VAS at postoperative day#1 | Postoperative day 1
  Maximum postoperative pain using the visual analogue scale

SECONDARY OUTCOMES:
Operation time | Time during operation
  Time spent during operation
Estimated blood loss | During operation
  Amount of blood loss during operation
Early postoperative complication | within 30 days from the operation
  Postoperative complications within 30 days from the operation
Hospital stay | Days until discharge
  Days until discharge
Time to first flatus | Days until first flatus
  Days until first flatus
Time to first soft fluid diet | Days until first soft fluid diet
  Days until first soft fluid diet
Maximum pain scores using VAS | From postoperative day 0 to 5
  Maximum pain scores using the visual analogue scale
EORTC-C30 and STO22 | Preoperative, 2 weeks after surgery, 1 month after surgery, 6 months after surgery, 12 months after surgery
  Quality of life questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hoon Ahn, M.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea